CLINICAL TRIAL: NCT06794606
Title: Multimodal Study for the Diagnosis and Treatment of Drug-resistant Focal Epilepsies
Brief Title: Study for the Diagnosis and Treatment of Drug-resistant Focal Epilepsies
Acronym: EpiBesta
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: EpiBesta
Record Dates: First submitted 2024-12-06; First posted 2025-01-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy
Keywords: Epilepsy surgery; drugs resistant focal epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — brain tissue, blood and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Epilepsy is a clinical condition that affects about fifty million people worldwide, with an estimated occurrence of 16-51 new cases per 100,000 people each year. In 60% of these patients, the origin of seizures is due to a localized (focal) alteration of the brain. In about 25 percent of patients with focal epilepsy, drug treatment is ineffective, a condition defined by the International League Against Epilepsy (ILAE) as drug-resistant epilepsy ; this condition results in a drastic reduction in quality of life associated with psychosocial dysfunction and an increased risk of sudden death. A possible treatment alternative for drug-resistant patients is ablation of the epileptogenic zone through surgical methods that are effective and safe when patients are carefully selected. The percentage of patients with epilepsy who are completely cured after surgery is about 70% for temporal lobe epilepsies, and can be as high as 90% in the case of some brain malformations.

Pre-surgical screening and therapeutic intervention (particularly surgery) have health care costs that are amortized over 2-6 years depending on the procedures required before surgery. In the last decade, moreover, the refinement of noninvasive/mini-invasive methods such as radiosurgery, Magnetic Resonance-guided Focused Ultrasound (MRgFUS) and laser interstitial thermal therapy (LiTT) have allowed us to hypothesize a possible specific treatment of drug-resistant patients with epileptogenic areas that are difficult to reach with traditional surgery and patients with complex comorbidities for whom the risks of standard resective surgery would outweigh the possible benefits. Finally, there is a subgroup of patients with drug-resistant epilepsy who cannot undergo ablative surgery. In these patients, seizures originate from multiple areas of the brain (multifocal epilepsy) or the epileptogenic area affects functionally eloquent areas. In these cases, alternative functional treatments are proposed, which aim to decrease the frequency and intensity of seizures and the need for medication, such as: i) application of a vagal stimulator, a pulse generator that is implanted in the chest and connected to the vagus nerve, ii) implantation of deep brain stimulation devices, iii) neuromodulation. Therefore, careful selection of patients during the diagnostic/pre-surgical process is crucial. The multimodal assessments under study, proposed in support of clinical practice, aim to improve such selection by analyzing the causative factors of seizures, the location of the epileptogenic zone, and the clinical-epileptological course of patients who are candidates for surgical or functional treatment of epilepsies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with focal epilepsy, long history of drug-resistant seizures, on mono- or polypharmacy antiepileptic therapy affected by known epileptogenic lesion or without lesions evident on neuroimaging investigations (cryptogenic). - - - Patients with recent onset of focal seizures, in mono- or polypharmacy, with controlled or rare seizures, or still in the absence of antiepileptic therapy affected by neoplastic lesion.

Exclusion Criteria:

* Patients in whom the diagnosis of epilepsy is doubtful. Patients with cognitive or psychiatric disorders that prevent participation in an interview, proper understanding of informed consent, or completion of questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with focal epilepsy, long history of drug-resistant seizures, on mono- or polypharmacy antiepileptic therapy affected by known epileptogenic lesion or without lesions evident on neuroimaging investigations (cryptogenic). - - Patients with recent onset of focal seizures, in mono- or polypharmacy, with controlled or rare seizures, or still in the absence of antiepileptic therapy affected by neoplastic lesion.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Treatment | 10 years
  To assess the clinical-epileptological course of patients with focal epilepsy who are candidates for surgical treatment of epilepsies
Alternative to resective surgery | 10 years
  To assess the clinical-epileptological course of patients with focal epilepsy who are candidates for diagnostic and therapeutic interventions as an alternative to conventional resective surgery.

SECONDARY OUTCOMES:
Investigate the factors | 10 years
  To investigate the factors (environmental/molecular/genetic) leading to the development of epilepsies, in particular the forms resistant to pharmacological treatment
Identify new approaches | 10 years
  To identify new and more effective non-invasive approaches in order to precisely identify the surgical target (epileptogenic zone) reducing the use of invasive monitoring and treatment techniques
Improving clinical outcomes | 10 years
  Improving clinical outcomes by reducing costs and risks associated with diagnostic and therapeutic procedures in epilepsy surgery
Database | 10 years
  Structuring a database of patients with drug-resistant focal epilepsy for future treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Carlo Besta Neurological Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No